CLINICAL TRIAL: NCT00710047
Title: A Randomised, Open-label, Single-centre, Crossover Study in Healthy Male Volunteers to Assess the Effect of Food on the Pharmacokinetics of a 10 mg Single Oral Dose of ZD4054 (Zibotentan)
Brief Title: Food Effect Study of a Single Dose of ZD4054 (Zibotentan)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Thomas Morris, BSc MB BCh MRCP FFPM, Medical Science Director, ZD4054, AstraZeneca R&D Alderely Park
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D4320C00028; ZD4054EudraCt 2008-002744-42
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2010-11

CONDITIONS: Healthy Volunteers
Keywords: ZD4054; Zibotentan; Healthy Volunteers
MeSH Terms: interventions — ZD4054

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Fasting state
  Interventions: Drug: ZD4054
- 2 (Experimental): after high-fat breakfast
  Interventions: Drug: ZD4054

INTERVENTIONS:
Drug: ZD4054 — one single 10mg dose
  Other Names: Zibotentan

SUMMARY:
The purpose of the study is to assess the effect of food on the pharmacokinetics of a 10 mg single oral dose of ZD4054 (Zibotentan)

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 and 30 kg/m2
* Medical and surgical history and physical examination without any clinically significant findings
* Able to consume standard FDA specified high-fat breakfast.

Exclusion Criteria:

* Definite or suspected personal history or family history of hypersensitivity to drugs that are endothelin antagonists; ie, ambrisentan, artrasentan, sitaxsetan and bosentan
* Medical diagnosis of migraine with an attack during the 12 months prior to Screening
* Use of prescription medication within 2 weeks before dosing

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
PK variables | frequent sampling occasions during study days

SECONDARY OUTCOMES:
Safety variables (adverse events, blood pressure, pulse, safety lab) | During the whole treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Morris, Study Director — AstraZeneca, Medical Science Director; David Wessels, Principal Investigator — Parexel
Locations (1):
- Research Site, Harrow, United Kingdom